CLINICAL TRIAL: NCT03529539
Title: Expanded Access for PSV Personalized Oncolytic Viruses
Acronym: PSV
Status: No longer available | Type: Expanded Access
Sponsor: EpicentRx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PSV
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: PSV

SUMMARY:
A compassionate use, expanded access protocol for patients who have exhausted all standard therapy having progressed on chemotherapy and immunotherapy.

DETAILED DESCRIPTION:
Patients will receive intratumoral or subcutaneous injection of an oncolytic virus called PSV (short for Personalized Virus) every other week until the occurrence of immune related RECIST progression, intolerable toxicity, change to another anti-cancer treatment due to lack of apparent benefit, or personal choice.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign a written informed consent form.
* Measurable or evaluable disease with least one (1) tumor that is accessible to intratumoral injection.
* Eastern Cooperative Group (ECOG) performance status is 0-3 at Screening.
* Acceptable liver function at Screening, as evidenced by:

  * Bilirubin ≤ 3.0 X upper limit of normal (ULN) since this patient has
  * been diagnosed with Gilbert's Disease
* AST (SGOT) and ALT (SGPT) ≤ 5 X ULN.
* Serum creatinine < 3 x institution upper limit of normal.
* Patient has acceptable hematologic status at Screening, as evidenced by:

  * Absolute neutrophil count ≥ 1,500 cells/mm3; and
  * Platelet count ≥ 70,000/mm3; and
  * Hemoglobin (HGB) ≥ 8.5 g/dL.
* Medically acceptable contraception.
* Willingness to comply with all protocol procedures, evaluations and rescue measures.

Exclusion Criteria:

* Presence of a serious co-morbid medical condition, or a clinically significant laboratory finding(s) that, in the opinion of the Investigator, suggests the presence of an infectious, endocrine, and/or other inadequately treated systemic disorder.
* An active bacterial, fungal, or viral infection.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: John Morris, MD, Principal Investigator — University of Cincinnati